CLINICAL TRIAL: NCT04002362
Title: Symptom Clusters in Children With Exacerbation-prone Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Anne M Fitzpatrick, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00111087; R01NR018666 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children
Keywords: Asthma; Pediatrics
MeSH Terms: conditions — Asthma | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Triamcinolone Acetonide (Experimental): Pediatric participants with exacerbation-prone asthma receiving an intramuscular injection of triamcinolone acetonide and are followed for 48 weeks.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — An intramuscular injection of triamcinolone acetonide (1 mg/kg, up to 40 mg maximum) is administered deep in the gluteal muscle by a trained registered nurse.
  Other Names: Kenalog

SUMMARY:
Pediatric participants with exacerbation-prone asthma will receive an intramuscular injection of triamcinolone acetonide and will be followed for 48 weeks. The study visit 2 weeks after the injection will assess the response to the study medication, while the remaining study visits will examine the temporal stability of the symptom clusters.

DETAILED DESCRIPTION:
Asthma symptom control is suboptimal in the majority of children in the United States, despite widespread availability of asthma controller medications and standardized treatment guidelines. While deaths from asthma have declined, 53.7% of children with asthma continue to experience an exacerbation each year and the associated public health burden is substantial.

While the factors responsible for poor asthma symptom control are complex and include limited access to care, poor adherence to preventative asthma medications, and exposures to environmental allergens and irritants such as tobacco smoke, it is also recognized that children with exacerbation-prone asthma are a heterogeneous group with differing clinical outcomes and longitudinal disease trajectories. Symptoms (defined as subjective sensations) can also be quite varied within and among affected children. Whereas some children have persistent, troublesome respiratory symptoms, others have respiratory symptoms only with upper respiratory infections. Mental health symptoms and social health symptoms have been inadequately characterized in this population, but some children with asthma also report depression and anxiety and impaired family functioning and relationships that may further worsen asthma outcomes. However, prior studies are limited by a narrow focus on individual symptoms in isolation. To date, there has been no attempt to identify symptom clusters (defined as two or more concurrent symptoms independent of other clusters) in children with exacerbation-prone asthma.

Poor understanding of symptom clusters is a major shortcoming in asthma symptom science. In other chronic disorders such as cancer, compared with a single symptom, symptom clusters of pain, fatigue, sleep disturbance and mood disturbance significantly worsen patient-reported outcomes of functional status and quality of life. There is also emerging evidence that interventions for one symptom within a cluster (i.e., cognitive-behavioral therapy for pain) reduce the severity of other symptoms within that cluster (i.e., fatigue and sleep disturbance). Because children with exacerbation-prone asthma rarely report a single symptom, greater knowledge of the assessment (and ultimately management) of symptom clusters in these children has the potential to significantly improve individualized treatment and clinical outcomes.

The researchers propose a 48-week cohort study to test the overarching hypothesis that symptom clusters and their associated inflammatory and metabolic pathways predict corticosteroid treatment responsiveness (primary objective outcome) and quality of life (patient-reported secondary outcome) in children 6- 21years of age with exacerbation-prone asthma. Participants will be given the option to either: 1) complete a single study visit, with telephone/email contacts and a review of their electronic medical record for up to 48 weeks after enrollment, or 2) complete the 48-week cohort study with scheduled study visits. Participants who select option 2 with follow-up over 48 weeks will also have the option to complete visits 3, 4 and 5 by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to less than 21 years at the enrollment visit
* Physician diagnosis of asthma
* History of an asthma exacerbation in the previous 12 months, defined as either:

  * Treatment with systemic corticosteroids, or
  * Increase in rescue medication use (i.e., albuterol or inhaled corticosteroid) for 24 hours or more, or
  * One or more missed school days due to asthma symptoms, or
  * An unscheduled visit for asthma at either a physician's office, urgent care, hospital emergency room, or
  * Hospitalization for asthma

Exclusion Criteria:

* Previous allergic reaction to systemic corticosteroids
* Hepatic, biliary, or renal disease that can interfere with drug metabolism/excretion
* Chronic medical disorders that may increase the risk of drug-related injury, including osteogenesis imperfecta (increased risk of fracture with corticosteroids), or Crohn's disease, ulcerative colitis, juvenile rheumatoid arthritis, clotting disorders, or Factor deficiency (increased risk of bleeding with corticosteroid therapy)
* Pregnancy
* Current smoking
* Congenital disorders or deformities of the chest wall, lungs or airways
* History of premature birth <35 weeks gestation
* Unwillingness to receive triamcinolone
* Planning to relocate before study completion

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fitzpatrick, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Altanta, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing three months following publication, with no end date.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the proposal. Proposals should be directed to anne.fitzpatrick@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Children's Center and Children's Healthcare of Atlanta in Atlanta, Georgia, USA. Participant enrollment began November 13, 2019 and all follow-up assessments for the Day 14 time point were completed by January 16, 2025. Follow-up assessments for the Week 48 time point were completed by December 24, 2025..
Period: Overall Study
Arm/Group | Triamcinolone Acetonide
Started | 68
Completed | 67
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Triamcinolone Acetonide: Pediatric participants with exacerbation-prone asthma receiving an intramuscular injection of triamcinolone acetonide and are followed for 48 weeks. An intramuscular injection of triamcinolone acetonide (1 mg/kg, up to 40 mg maximum) is administered deep in the gluteal muscle by a trained registered nurse.
Arm/Group | Triamcinolone Acetonide
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 50
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Questionnaire (ACQ) Score
Description: Responsiveness to the study treatment is assessed with the Asthma Control Questionnaire (ACQ). This 7-item questionnaire includes questions related to daytime and nocturnal symptoms, short-acting bronchodilator use, and lung function during the clinic visit on that day. Participants report how difficult their asthma was to control on a scale from 0 (no impairment) to 6 (maximum impairment). Total raw scores range from 0 to 42, with higher scores indicating poorer asthma control. Responsiveness to treatment is determined with the mean difference in ACQ score the baseline visit and the Day 14 visit, with a reduction of 0.5 considered a minimally important difference.
Time Frame: Baseline, Day 14
Population: This analysis includes participants who completed both the Baseline and Day 14 study assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone Acetonide
Number analyzed (Participants) | 67
score on a scale | 0.52 (0.89)

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Asthma Impact Scale (PAIS)
Description: Quality of life is assessed with the 8-item PAIS instrument. As with all PROMIS measures, the PAIS is scored on the T-score metric, with higher scores reflecting more of the concept being measured. On the T-score metric, 50 is the mean of the reference population and 10 is the standard deviation, thus, scores of 40 and 60 are one standard deviation lower and higher than the mean of the reference population, respectively.
Time Frame: Weeks 16, 32, and 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone Acetonide
Number analyzed (Participants) | 62
score on a scale
  Week 16 | 42.7 (9.8)
  Week 32 | 42.9 (9.8)
  Week 48 | 44.7 (10.7)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of enrollment and continued through the Day 14 assessment, for a total of 14 days.
Arm/Group | Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04002362/Prot_SAP_001.pdf
  • Informed Consent Form (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04002362/ICF_000.pdf